CLINICAL TRIAL: NCT06445114
Title: ULTRA-HPV Using Circulating Tumor DNA to Risk Adapt Post-operative Therapy for HPV Associated Oropharyngeal Cancer
Brief Title: Using CircuLating Tumor DNA to Risk Adapt Post-Operative Therapy for HPV-associated Oropharyngeal Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Zachary Zumsteg (Other)
Responsible Party: Sponsor-Investigator, Zachary Zumsteg, Sponsor-Investigator, Cedars-Sinai Medical Center
Organization: Cedars-Sinai Medical Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IIT2023-14-ZUMSTEG-ULTRA-HPV
Record Dates: First submitted 2024-05-22; First posted 2024-06-06 (Actual); Last update posted 2025-11-04 (Actual); Status verified 2025-11

CONDITIONS: Oropharyngeal Cancer; Carcinoma
Keywords: Transoral Robotic Surgery (TORS); pT0 tumors (unknown primary); p16
MeSH Terms: conditions — Oropharyngeal Neoplasms; Carcinoma | interventions — Cisplatin; Chemoradiotherapy

STUDY DESIGN:
Intervention Model Description: Prospective single arm multicenter clinical trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Single Arm (Experimental): Low risk pathology with post-op HPV DNA (-): cisplatin-based chemoradiation with 30 Gy in 15 fractions and 3 cycles of weekly cisplatin 40mg/m2 IV on Days 1, 8, and 15 of radiation.
  Low risk pathology with post-op HPV DNA (+): cisplatin-based chemoradiation with 40 Gy in 20 fractions and 4 cycles of weekly cisplatin 40mg/m2 IV on Days 1, 8, 15, and 22 of radiation.
  High risk pathology with post-op HPV DNA (-), excluding patients with both 5 LN+ and ENE+ or pre-op HPV DNA≤12 copies/mL: cisplatin-based radiation with 40 Gy in 20 fractions and 4 cycles of weekly cisplatin 40mg/m2 IV on Days 1, 8, 15, and 22 of radiation.
  High risk pathology with post-op HPV DNA (+) OR pre-op HPV DNA≤12 copies/mL OR both 5 or more LN+ and ENE+: cisplatin-based radiation with 50 Gy in 25 fractions with 5 cycles of weekly cisplatin 40mg/m2 IV on Days 1, 8, 15, 22, and 29 of radiation.
  Interventions: Drug: Cisplatin

INTERVENTIONS:
Drug: Cisplatin — Low risk pathology with post-op HPV DNA (-): cisplatin-based chemoradiation with 30 Gy in 15 fractions and 3 cycles of weekly cisplatin 40mg/m2 IV on Days 1, 8, and 15 of radiation.
  Low risk pathology with post-op HPV DNA (+): cisplatin-based chemoradiation with 40 Gy in 20 fractions and 4 cycles of weekly cisplatin 40mg/m2 IV on Days 1, 8, 15, and 22 of radiation.
  High risk pathology with post-op HPV DNA (-), excluding patients with both 5 LN+ and ENE+ or pre-op HPV DNA≤12 copies/mL: cisplatin-based radiation with 40 Gy in 20 fractions and 4 cycles of weekly cisplatin 40mg/m2 IV on Days 1, 8, 15, and 22 of radiation.
  High risk pathology with post-op HPV DNA (+) OR pre-op HPV DNA≤12 copies/mL OR both 5 or more LN+ and ENE+: cisplatin-based radiation with 50 Gy in 25 fractions with 5 cycles of weekly cisplatin 40mg/m2 IV on Days 1, 8, 15, 22, and 29 of radiation.
  Other Names: Chemoradiation

SUMMARY:
This is a single institution phase II study that will enroll patients with T0-3N0-2 p16-positive oropharyngeal squamous cell carcinoma (OSCC) undergoing resection of all gross visible disease at the primary site and in the lymph nodes.

DETAILED DESCRIPTION:
All eligible patients will be treated with a de-intensified cisplatin-based chemoradiation regimen after undergoing transoral robotic surgery. Enrolled patients will be risk-assessed and assigned to specific regimens based on a combination of their post-operative cTTMV-HPV DNA, as determined by results from NavDx kits by Naveris, and pathologic features. All patients will receive a dose of 40 mg/m2 IV weekly concurrently with radiation therapy. Patients ineligible to receive cisplatin at this dose will undergo modified sydtemic therapy. Patients will recieve concurrent radiation in a dose of 30 Gy in 15 fractions to the primary tumor bed, ipsilateral neck +/- contralateral neck. Based on risk-stratification, some patients will receive a sequential boost of 10 Gy over 5 fractions or 20 Gy over 10 fractions.

ELIGIBILITY:
Inclusion Criteria:

* AJCC 8th edition T0-3N0-2 p16-positive oropharyngeal (tonsil, base of tongue, glossotonsillar sulcus, soft palate, oropharyngeal wall) squamous cell carcinoma or squamous cell carcinoma of unknown primary involving the cervical lymph nodes. Cytologic diagnosis from a cervical lymph node is sufficient for diagnosis in the presence of clinical evidence of a primary tumor in the oropharynx.
* For patients with pT0 tumors (unknown primary), there must be at least one metastatic lymph node present in cervical level II.
* p16 is strongly positive by immunohistochemistry or high-risk HPV is detected by in-situ hybridization.
* Have undergone or will undergo gross total resection of all known disease in the head and neck via transoral robotic surgery. For patients with clinical unknown primary tumors, a patient must undergo both ipsilateral tonsillectomy and base of tongue resection unless the primary is identified clinically or pathologically at the time of surgery. If the primary is identified, then only resection of the primary site is required. If the primary tumor is resected with negative margins with a non-robotic surgery, such as a diagnostic tonsillectomy, this is considered acceptable and further robotic surgery is not necessary.
* Have undergone or will undergo neck dissection.
* Have at least one of the following after surgery:

  * Pathologic stage T3
  * 2 or more positive lymph nodes
  * At least one lymph node >3cm
  * Contralateral lymph node involvement
  * Lymphovascular invasion
  * Perineural invasion
  * Extranodal extension
  * Close/positive margins: Close margins are considered ≤3mm from the peripheral margins and ≤1mm from the deep margin on the en bloc specimen, unless the area of close margin is re-resected and without carcinoma.
* Patients consented preoperatively are required to have detectable cTTMV-HPV DNA based on pre-operative NavDx testing. For patients consented post-operatively, NavDx testing should be performed on the tumor tissue to ensure detectable HPV DNA and for HPV subtyping.
* Age ≥ 18 years old
* ECOG performance status 0 or 2 within 56 days of start of chemoradiation.
* Women of childbearing potential require a negative serum or urine pregnancy test within 28 days prior to start of chemoradiation.
* Written informed consent obtained from subject and ability for subject to comply with the requirements of the study.
* Adequate hematologic and renal function within 56 days of start of chemoradiation, defined as:

  * Hemoglobin ≥ 9.0 g/dL
  * Platelets ≥ 100, 000 cells/mm3
  * ANC ≥ 1.5 X 109/L
  * Total bilirubin ≤ 1.5 x upper limit of normal (ULN)
  * Aspartate aminotransferase/alanine aminotransferase ≤ 3.0 x upper limit of normal (ULN)
  * Serum creatinine ≤1.5 x upper limit of normal (ULN) OR a calculated creatinine clearance ≥50 mL/min estimated using the following Cockcroft-Gault equation

Exclusion Criteria:

* AJCC 8th edition pT4 or cN3 disease.
* Radiologic or clinical evidence of distant metastasis.
* Recurrent disease.
* Inability to achieve gross total resection at time of surgery.
* Greater than 56 days (8 weeks) after surgical resection of the primary site.
* Prior radiation to the head and neck > 30 Gy.
* Prior active invasive (not in situ) malignancy within the prior 2 years, excluding cutaneous basal cell or squamous cell carcinoma, low or intermediate risk prostate cancer, papillary thyroid cancer, stage T1aN0 kidney cancer, low-grade T1-2N0 salivary cancer, AJCC 8th edition stage I-II breast cancer, well-differentiated neuroendocrine tumors (e.g., carcinoid tumors), low grade non-Hodgkin lymphoma, or Stage 0, I, and III cutaneous melanomas. Patients with synchronous or multifocal oropharyngeal cancers are not excluded, as long as at least one of these tumors meet inclusion criteria for the trial.
* Severe, active co-morbidity, defined as follows:

  * Unstable angina and/or congestive heart failure requiring hospitalization within the last 6 months
  * Transmural myocardial infarction within the last 6 months
  * Acute bacterial or fungal infection requiring intravenous antibiotics at the time of enrollment
  * Hepatic insufficiency resulting in clinical jaundice and/or known coagulation defects
* Moderate to severe hearing loss.
* Active connective tissue disease (e.g. systemic lupus erythematous, scleroderma) requiring immunosuppression.
* Pregnant or breast-feeding women.
* Prior allergic reaction to cisplatin.
* Live vaccines within 30 days prior to the first dose of chemoradiation. Examples of live vaccines include, but are not limited to, the following: measles, mumps, rubella, chicken pox, yellow fever, rabies, BCG, and typhoid (oral vaccine). Season influenza vaccines for injection are generally killed virus vaccines and are allowed; however intranasal influenza vaccines (e.g. Flu-Mist®) are live attenuated vaccines and are not allowed.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-05-12 (Actual); Primary Completion 2032-06 (Estimated); Study Completion 2032-06 (Estimated)

PRIMARY OUTCOMES:
2-year progression-free (PFS) | 2 Years
  The primary objective of this study is to assess the 2-year progression-free survival (PFS) of de-intensified post-operative chemoradiation in patients with HPV-associated oropharyngeal cancer when basing treatment intensity on both standard pathologic features and post-operative Blood-based circulating tumor tissue modified viral (cTTMV-HPV DNA)

SECONDARY OUTCOMES:
Overall Survival (OS) | 2 Years
  Proportion of patients alive, based on time from enrollment to death from any cause.
Locoregional Control | 2 Years
  Proportion of patients without local recurrence or regional recurrence, as defined above, based on the time from enrollment to the first evidence of either local or regional recurrence, irrespective of prior distant recurrence. Death from causes unrelated to cancer is a competing event.
Distant Control | 2 Years
  Proportion of patients without distant recurrence, based on time from enrollment to distant recurrence, irrespective of prior local or regional recurrence. Distant metastasis includes any recurrent disease outside of the head and neck, cervical lymph nodes, or retropharyngeal lymph nodes. Death from causes unrelated to cancer is a competing event.
Cause-Specific Survival | 2 Years
  Proportion of patients without oropharyngeal cancer-related or treatment-related death, based on time from enrollment to death from oropharyngeal cancer or treatment. Death from other causes is a competing event.
Mean change in patient-reported outcomes using Patient-Reported Outcomes Version of the Common Terminology Criteria for Adverse Events (PRO-CTCAE) | 2 Years
  To assess quality of life changes before, during and after treatment via Patient-Reported Outcomes Version of the Common Terminology Criteria for Adverse Events (PRO-CTCAE)
  PRO-CTCAE responses are scored from 0 to 4 (or 0/1 for absent/present), with lower scoring indicating an absence of symptoms to higher scoring reflecting higher severity of symptoms.
Mean change in patient-reported outcomes using Hearing Handicap Inventory for Adults (HHIA-S) | 2 Years
  To assess quality of life changes before, during and after treatment via Hearing Handicap Inventory for Adults (HHIA-S). The scale ranges from 0 to 4 (0 - no, 2 - sometimes, 4- yes) for each question identifying problems with hearing loss, as self-reported by patients. The total number of points for the 25 questions range from 0 to 100, with 0 indicating no handicap to 100 indicating total handicap.
Mean change in patient-reported outcomes using European Organisation for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire (QLQ-C30) | 2 Years
  To assess quality of life changes before, during and after treatment via EORTC QLQ-C30. The EORTC QLQ-C30 is composed of both multi-item scales and single-item measures. These include 5 functional scales, 3 symptom scales, a global health status / QoL, and 6 single items. All of the scales and single-item measures range in score from 0-100. A high scale score represents a higher response level and represents a high/healthy level of functioning, a high score for the global health status/QoL represents a high QoL, but a high score for a symptom scale represents a high level of problems. Most questions are scored 1 to 4, with exception to global health questions scored from 1 to 7. The raw scores are then standardized by a linear transformation, so that scores range from 0 to 100; a higher score represents a higher ("better") level of functioning, or a higher ("worse") level of symptoms.
Mean change in patient-reported outcomes using the MD Anderson Dysphagia Inventory (MDADI) | 2 Years
  To assess quality of life changes before, during and after treatment via the MD Anderson Dysphagia Index (MDADI). The MDADI is a patient-reported, 20-item scale that quantifies four domains: an individual's global (G), physical (P), emotional (E), and functional (F) perceptions of their swallowing ability. Two summary scores can be obtained from the MDADI: 1) global and 2) composite. The global scale is a single question, scored individually, to assess the overall impact that swallowing abilities have on quality of life. The composite MDADI score summarizes overall performance on remaining 19-items of the MDADI, as a weighted average of the physical, emotional, and functional subscale questions. Summary and subscale MDADI scores are normalized to range from 20 (extremely low functioning) to 100 (high functioning). Five possible responses to the items on the MDADI are: strongly agree, agree, no opinion, disagree, and strongly disagree, and scored on a scale of 1 to 5 respectively.
Mean change in patient-reported outcomes using University of Michigan Xerostomia-Related Quality of Life Scale (XeQoLS) | 2 Years
  To assess quality of life changes before, during and after treatment via the University of Michigan Xerostomia-Related Quality of Life Scale (XeQoLS). XeQOLS is a patient-reported, 15-item scale that measures four domains: physical functioning, pain/discomfort, personal/psychologic functioning, and social functioning. Patient responses to all four domains are averaged, and the total scores range from 0 to 4; an increased xerostomia burden is indicated by a higher score.
Mean change in patient-reported outcomes using 5-level version of the EuroQol five dimensional instrument EQ-5D-5L | 2 Years
  To assess quality of life changes before, during and after treatment via the 5-level version of the EuroQol five dimensional instrument EQ-5D-5L.The EQ-5D-5L descriptive system comprises of five dimensions: (MOBILITY, SELF-CARE, USUAL ACTIVITIES, PAIN / DISCOMFORT and ANXIETY / DEPRESSION), with each dimension having five response levels: no problems, slight problems, moderate problems, severe problems, unable to /extreme problems - severity level of each dimension are coded from 1 to 5, respectively. The visual analog scale (EQ VAS) attached to this questionnaire records the respondent's overall self-rated perception of current health status on a vertical visual analogue scale, where the endpoints are scored from 0 to 100, 100 being the 'The best health you can imagine' and 0 indicating 'The worst health you can imagine'
Mean change in Dysphagia using MDADI | 2 Years
  To assess dysphagia before, during, and after treatment with the MD Anderson Dysphagia Inventory (MDADI) tool. The MDADI is a patient-reported, 20-item scale that quantifies four domains: an individual's global (G), physical (P), emotional (E), and functional (F) perceptions of their swallowing ability. Two summary scores can be obtained from the MDADI: 1) global and 2) composite. The global scale is a single question, scored individually, to assess the overall impact that swallowing abilities have on quality of life. The composite MDADI score summarizes overall performance on remaining 19-items of the MDADI, as a weighted average of the physical, emotional, and functional subscale questions. Summary and subscale MDADI scores are normalized to range from 20 (extremely low functioning) to 100 (high functioning). Five possible responses to the items on the MDADI are: strongly agree, agree, no opinion, disagree, and strongly disagree, and scored on a scale of 1 to 5 respectively.
Mean change in Dysphagia using Modified Barium Swallow | 2 Years
  To assess dysphagia before, during, and after treatment with the modified barium swallow. MBS is an analysis of swallowing through three phases: oral (mouth), pharyngeal (throat) and upper esophagus. A Modified Barium Swallow Study (MBSS) is a special x-ray that allows the Radiologist (who specializes in using x-rays) and Speech Language Pathologist (SLP) to identify why you are having trouble swallowing. The MBS provides quantitative evaluation of 17 physiologic components of swallowing distributed across three functional domains: oral, pharyngeal, and esophageal. MBS components are scored on an ordinal scale from 0 (indicating no impairment) to a maximum of 2, 3, or 4, depending on the specific component.
2-year Progression-Free Survival | 2 Years
  To assess the 2-year PFS (Progression-Free Survival) in the high-risk [extranodal extension (ENE), positive margins, ≥5 positive lymph nodes (LNs)] and intermediate-risk [T3, close margins, LN size > 3cm, 2 or more LN+, lymphovascular invasion (LVI), perineural invasion (PNI)] subgroups separately. The difference between the proportion of patients alive and without evidence of local, regional, or distant recurrence at 2 years from study enrollment, in high-risk and intermediate subgroups.

CONTACTS AND LOCATIONS:
Overall Officials: Zachary S Zumsteg, MD, Principal Investigator — Cedars-Sinai Medical Center
Locations (4):
- United States (4):
  - Cedars-Sinai Cancer at Beverly Hills (THO), Beverly Hills, California
  - Cedars Sinai Medical Center, Los Angeles, California
  - CS Cancer at Valley Oncology Medical Group, Tarzana, California
  - CS Cancer at the Hunt Cancer Center, Torrance, California

IPD SHARING:
Plan to Share IPD: No